CLINICAL TRIAL: NCT02849132
Title: Effect of Entecavir Treatment on Regression and Long-term Disease Outcome in Patients With HBV-induced Liver Fibrosis and Cirrhosis (Regress Extension Study)
Brief Title: Effect of Entecavir Treatment on Regression and Disease Outcome in HBV-induced Liver Fibrosis and Cirrhosis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Peking University People's Hospital (Other); Fudan University (Other); Affiliated Hospital of Yanbian University (Unknown); Shanghai Public Health Clinical Center (Other Government); Beijing YouAn Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaojuan Ou, Vice-Director of Liver Research Center, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016ZX10002011
Record Dates: First submitted 2016-07-22; First posted 2016-07-29 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis B; Liver Cirrhosis
MeSH Terms: conditions — Hepatitis B; Liver Cirrhosis | interventions — entecavir

ARMS (1):
- Treatment group (Experimental): entecavir oral，0.5mg daily for 8 years
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — oral entecavir 0.5mg daily for 8 years

SUMMARY:
Patients who have completed 2 years follow-up of the past National 12th Five-Year Major Project on Infectious Diseases will receive another 8 years treatment with entecavir (10 years in total). Collect serology, imaging, and other clinical data to evaluate the incidence and mortality of decompensated cirrhosis and hepatocellular carcinoma. Understand the effects of long-term antiviral therapy on HBV-induced liver fibrosis/cirrhosis.

DETAILED DESCRIPTION:
Patients who have completed 2-years entecavir-based treatment in Regress Study will receive another 8 years of entecavir extension therapy. Patients will be assessed at baseline and every six months for blood cell count, liver function test, HBV-DNA, AFP, prothrombin time, liver ultrasonography, and Fibroscan; A third liver biopsy will be performed at the 5th year of treatment in patients who have significant fibrosis at second biopsy. CT /MRI and endoscopy will be performed at baseline and the 5th and 10th year of treatment.

ELIGIBILITY:
Inclusion Criteria:

- Subjects who completed the 2 years of entecavir-based therapy in Regress study; Subjects who are willing to participate the extension study.

Exclusion Criteria:

- Any complication of severe heart, lung, kidney, brain, blood diseases or other important systematic diseases; Pregnant women; Subjects who could not compliance with the protocol judged by investigators; Subjects who are not suitable for the study judged by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Fibrosis regression rate | year 3
  Ishak fibrosis score decrease after long-term treatment
Cumulative incidence of liver decompensation | year 8
  Cumulative incidence of liver decompensation (including ascites, hepatic encephalopathy, esophageal varices bleeding and Hepatocellular Carcinoma) and death after long-term treatment

SECONDARY OUTCOMES:
Virological response | year 3, 5, 7 and 10
  Percentage of patients achieving hepatitis B virus (HBV) DNA < 20IU/mL at year 3, 5, 7 and 10
Aminotransferase response | year 3, 5, 7 and 10
  The percentage of patients with alanine aminotransferase (ALT) normalization at year 3, 5, 7 and 10
HBeAg loss or HBeAg seroconversion | year 2, 5, 7 and 10
  Percentage of patients with HBeAg loss or HBeAg seroconversion at year 2, 5, 7 and 10
HBsAg loss or HBsAg seroconversion rate | year 2, 5, 7 and 10
  Percentage of patients with HBsAg loss or HBsAg seroconversion at year 2, 5, 7 and 10
Dynamic changes of Child-Pugh score | year 3, 5, 7 and 10
  Dynamic changes of Child-Pugh score after 3, 5, 7 and 10 years of treatment
Dynamic changes of MELD score | year 3, 5, 7 and 10
  Dynamic changes of MELD score after 3, 5, 7 and 10 years of treatment
Dynamic changes of liver stiffness values measured by Transient Elastography | year 3, 5, 7 and 10
  Dynamic changes of liver stiffness values after 3, 5, 7 and 10 years of treatment
Improvement of life quality (SF36 and EQ-5D) | year 3, 5, 7 and 10
  Improvement of life quality after 3, 5, 7 and 10 years of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojuan Ou, Principal Investigator — Beijing Friendship Hospital
Locations (20):
- China (20):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - 302 Military Hospital Of China, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - NanfangHospital,Southern Medical University, Guangzhou, Guangdong
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Shijiazhuang Fifth Hospital, Shijiazhuang, Hebei
  - Tongji Hospital, Tongji Medical College , Huazhong University of Science and Technology, Wuhan, Hubei
  - The Affiliated Hospital of Yanbian University, Yanji, Jilin
  - Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xijing Hospital, Fourth Military Medical University, Xi’an, Shanxi
  - Tianjin Xiqing Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Tianjin Third Central Hospital, Tianjin

REFERENCES:
- [Background] Arvaniti V, D'Amico G, Fede G, Manousou P, Tsochatzis E, Pleguezuelo M, Burroughs AK. Infections in patients with cirrhosis increase mortality four-fold and should be used in determining prognosis. Gastroenterology. 2010 Oct;139(4):1246-56, 1256.e1-5. doi: 10.1053/j.gastro.2010.06.019. Epub 2010 Jun 14. PMID 20558165
- [Background] Liaw YF, Sung JJ, Chow WC, Farrell G, Lee CZ, Yuen H, Tanwandee T, Tao QM, Shue K, Keene ON, Dixon JS, Gray DF, Sabbat J; Cirrhosis Asian Lamivudine Multicentre Study Group. Lamivudine for patients with chronic hepatitis B and advanced liver disease. N Engl J Med. 2004 Oct 7;351(15):1521-31. doi: 10.1056/NEJMoa033364. PMID 15470215
- [Derived] Zhang J, Chen S, Zhou J, Wang B, Wu X, Xu X, Zhao X, Kong Y, Ou X, Sun Y, You H. Serial Liver Stiffness Measurement and Serum Biomarkers Are Not Strong Predictors of the Regression of Fibrosis among Chronic Hepatitis B Patients Receiving Antiviral Therapy Based on Triple Liver Biopsies. Gut Liver. 2025 Nov 15;19(6):889-899. doi: 10.5009/gnl250008. PMID 41234032
- [Derived] Wu X, Hong J, Zhou J, Sun Y, Li L, Xie W, Piao H, Xu X, Jiang W, Feng B, Chen Y, Xu M, Cheng J, Meng T, Wang B, Chen S, Kong Y, Ou X, You H, Jia J. Health-related quality of life improves after entecavir treatment in patients with compensated HBV cirrhosis. Hepatol Int. 2021 Dec;15(6):1318-1327. doi: 10.1007/s12072-021-10240-4. Epub 2021 Nov 29. PMID 34843068
- [Derived] Wu X, Zhou J, Sun Y, Ding H, Chen G, Xie W, Piao H, Xu X, Jiang W, Ma H, Ma A, Chen Y, Xu M, Cheng J, Xu Y, Meng T, Wang B, Chen S, Shi Y, Kong Y, Ou X, You H, Jia J. Prediction of liver-related events in patients with compensated HBV-induced cirrhosis receiving antiviral therapy. Hepatol Int. 2021 Feb;15(1):82-92. doi: 10.1007/s12072-020-10114-1. Epub 2021 Jan 18. PMID 33460002
- [Derived] Yang JM, Chen LP, Wang YJ, Lyu B, Zhao H, Shang ZY, Li J, Fan ZY, Wu SD, Ming X, Li X, Huang SP, Cheng JL. Entecavir add-on Peg-interferon therapy plays a positive role in reversing hepatic fibrosis in treatment-naive chronic hepatitis B patients: a prospective and randomized controlled trial. Chin Med J (Engl). 2020 Jul 20;133(14):1639-1648. doi: 10.1097/CM9.0000000000000857. PMID 32568867